CLINICAL TRIAL: NCT03258944
Title: Breath-Stacking and Ventilatory Muscle Strength
Brief Title: Ventilatory Muscle Training by Breath-Stacking in Healthy Youngsters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, PhD, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VMTBS- HY
Record Dates: First submitted 2017-07-21; First posted 2017-08-23 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breath-Stacking (Experimental): Participants will be seated, with their elbows resting on the table, holding the face mask attached to a T-tube and a one-way valve. They will be instructed to inspire and force the expiration inside the mask. The training will be conducted three times a week for a period of four weeks, totaling twelve sessions. The breath-stacking application protocol will consist of three three-minute series, with a three-minute recovery interval between each series, obtaining a total time of fifteen minutes in each session
  Interventions: Other: Breath-Stacking

INTERVENTIONS:
Other: Breath-Stacking — Participants will be seated, with their elbows resting on the table, holding the face mask attached to a T-tube and a one-way valve. They will be instructed to inspire and force the expiration inside the mask. The training will be conducted three times a week for a period of four weeks, totaling twelve sessions. The breath-stacking application protocol will consist of three three-minute series, with a three-minute recovery interval between each series, obtaining a total time of fifteen minutes in each session.

SUMMARY:
In several diseases in which muscle weakness is a determining factor for morbidity and mortality, inspiratory muscle training has been shown to be useful in improving the function of ventilatory muscles, delaying or minimizing the development of complications due to the reduction of inspiratory muscle strength.

The breath-stacking technique emerges as an easily applicable alternative, and it can be used in poorly collaborative patients. The technique described in the literature aims to increase pulmonary volumes.

This gain occurs with the coupling of a silicone mask on the patient's face, a unidirectional valve and with the expiratory branch occluded. Thus, inspirations occur sequentially in this medium, generating pulmonary hyperinflation and increasing the contractility power of the expiratory muscles, which are fundamental for coughing. This hyperinflation also improves the peripheral air distribution in the lungs by increasing intrathoracic pressure.

The objective of this study is to evaluate the effect of the breath-stacking (BS) technique on the ventilatory muscle strength of young and healthy individuals.

DETAILED DESCRIPTION:
Initially, participants will be submitted to a learning session on the evaluation of ventilatory muscle strength and the breath-stacking technique. Between 24-72 hours after the learning, the evaluation of the muscular muscular strength will be performed through the maximal inspiratory pressure (MIP) and the maximum expiratory pressure (MEP). PI max will be measured from a maximum expiration; While PE max will be measured from a maximum inspiration, using a digital manovacuometer (MVD 300®)

ELIGIBILITY:
Inclusion Criteria:

* No signs and symptoms of pulmonary diseases, normal ventilatory muscle strength and agreement to participate and sign the informed consent form.

Exclusion Criteria:

* Presenting neuromuscular diseases, claustrophobia, ruptured eardrum, history of spontaneous pneumothorax and playing wind instruments or being a singer. Sample loss will be considered as non-attendance at all training sessions.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Ventilatory Muscle Strength | four weeks
  Maximum inspiratory and expiratory pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No